## Straumann BLT CIR-ECL-2016-03 STATISTICAL ANALYSIS

Study Number: CIR-ECL-2016-03

Protocol Version: 1.2 Version Date: 07/06/2017

**Department:** Oral and Maxillofacial Surgery

Research Line: Oral Invalidity

**Research Title:** Evaluation of marginal bone loss in Straumann® BLT implants in patients with posterior partial edentulism. A randomized clinical study comparing direct implant

connection vs. intermediate abutment.

## 1. OBJECTIVES

The primary objective of the study is to compare the radiographic evolution of implants between two surgical techniques: direct connection vs. intermediate abutment.

## 2. SAMPLE AND STATISTICAL METHODOLOGY

The study sample consists of 30 patients undergoing rehabilitation with implants in two posterior sector positions. The group includes 22 men (73.3%) and 8 women (26.7%), divided into two groups according to the applied technique:

- **Direct connection group (control):** n=12 patients
- **Intermediate abutment group (test):** n=18 patients

The test group is further subdivided into two subgroups based on abutment height:

- **Subgroup H1 mm:** n=7 patients
- **Subgroup H2.5 mm:** n=11 patients

Since each patient contributes two implants (mesial and distal) to the study, the previous figures are doubled at the implant level, totaling 60 implants:

- **Direct connection group (control):** n=24 implants
- **Intermediate abutment group (test):** n=36 implants
- **Subgroup H1 mm:** n=14 implants
- **Subgroup H2.5 mm:** n=22 implants

The study design corresponds to an RCT with multilevel data: patient and implant.

The study collects **bone level (BL) measurements** in the mesial and distal areas of each implant at different time points:

- T1 (surgery)
- T2 (crowns placement)
- T3 (4 months)
- T4 (6 months)
- T5 (12 months)
- T6 (24 months)

Bone loss (MBL) at each time point Tj is calculated as the difference between T1 and Tj, following the investigator's database example:

Example: MBL T1T6 = BL T1 - BL T6.

Descriptive analysis provides key statistics for all variables collected in the study: absolute and relative frequencies (for categorical variables) and mean, standard deviation, range, median, and quartiles (for continuous variables). A complete report of this analysis is available in an appendix, presented in table format.

The radiographic variables **BL** and **MBL** are described for each zone (mesial and distal) of each implant (mesial and distal) and also averaged for mesial implants, distal implants, and total implants (mean of both).

A **Shapiro-Wilk test** was conducted to verify the normal distribution of **MBL** across different time points and within each group, yielding a confirmatory result (**p>0.05**).

## **Inferential Analysis**

To study the dependent variable MBL, linear models under the GEE (Generalized Estimating Equations) approach are applied to assess mean differences by group. Beta coefficient estimates with 95% confidence intervals (CIs) are obtained using the Wald Chi-square statistic.

The **GEE analysis methodology** is justified due to the intra-subject correlation inherent in the multi-level data structure (patients contribute multiple implants to the study).

The **same GEE methodology** is used to examine the effect of **intermediate abutment height** within the test group.

Similar linear models were applied to evaluate **overall bone loss progression** over the follow-up period and to analyze potential differences between mesial and distal implant positions or between mesial and distal areas within an implant.

Conventional association tests (Chi-square, Fisher's exact test) were used at the patient level to assess the homogeneity of the test and control groups.

The significance level used in the analyses was 5% ( $\alpha=0.05$ ).

A general linear model as described achieves 70% power to detect a mean MBL difference corresponding to a large effect size (d=0.8) between groups with 95% confidence. This power accounts for the dependency between observations, assuming a total of 60 implants in 30 different patients and a moderate intra-class correlation (ICC=0.5).